CLINICAL TRIAL: NCT00038909
Title: Factor VIII Mutation Testing Program in Previously Untreated Patients (PUPs) With Hemophilia A Participating in ReFacto® Study
Brief Title: Study Evaluating ReFacto in Hemophilia A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 3082A1-302
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

INTERVENTIONS:
Drug: BDDrFVII

SUMMARY:
To identify the causative mutations in previously untreated patients with hemophilia A enrolled in the ReFacto® clinical safety and efficacy study CTN 93-R833-0XX/C9741-28, using two established hemophilia mutation testing laboratories (one in Europe and one in North America).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were or are enrolled in Study CTN 93-R833-0XX/C9741-28, and have been treated with ReFacto® during this study are eligible for participation.
* The patient (or legal guardian) must be willing to give written informed consent before any study-related procedures are performed.
* A blood sample will be collected from each patient for the purpose of this study and will be analyzed at one or both of the designated central laboratories.

Exclusion Criteria:

* Any condition which, in the investigator's opinion, places the patient at undue risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 1994-09; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer